CLINICAL TRIAL: NCT04260906
Title: The Impact Of Auricular Vagus Nerve Stimulation On Pain And Life Quality In Patients With Fibromyalgia Syndrome
Brief Title: Auricular Vagus Nerve Stimulation For Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, hasan kerem alptekin, director of health sciences institute, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vagusstim
Record Dates: First submitted 2020-02-03; First posted 2020-02-07 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia; Myofascial Pain Syndrome
Keywords: Fibromyalgia Syndrome; Auricular Vagus Nerve Stimulation
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve stimulation (Active Comparator): Patients were admitted to the treatment as day visitors. Vagus nerve stimulation is carried out with a TENS device, which has specially designed surface electrodes in the shape of earphones, the size of which can be selected according to ear size. Electrodes were placed to correspond with the inner and rear surfaces of the tragus and the concha for both ears . The application is carried out, for 30 minutes, using a biphasic, asymmetrical waveform with a pulse duration that is less than 500 microseconds and a frequency of 10 Hertz.
  Interventions: Device: Vagus nerve stimulator
- exercise (Active Comparator): The exercise group was assigned a program, which consisted of strengthening, stretching, isometric and posture exercises, targeting the body and upper and lower extremities. That program was home-based and the program was requested to be completed. Patients were asked to attend weekly face to face sessions with a total of 4 of these sessions in the study duration.
  Interventions: Other: exercise

INTERVENTIONS:
Device: Vagus nerve stimulator — Vagus nerve stimulation is carried out with a TENS device, which has specially designed surface electrodes in the shape of earphones, the size of which can be selected according to ear size. Electrodes were placed to correspond with the inner and rear surfaces of the tragus and the concha for both ears (Figure 1). The application is carried out, for 30 minutes, using a biphasic, asymmetrical waveform with a pulse duration that is less than 500 microseconds and a frequency of 10 Hertz.
  Arms: Vagus nerve stimulation
Other: exercise — The exercise group was assigned a program, which consisted of strengthening, stretching, isometric and posture exercises, targeting the body and upper and lower extremities. That program was home-based and the program was requested to be completed. Patients were asked to attend weekly face to face sessions with a total of 4 of these sessions in the study duration.
  Arms: exercise

SUMMARY:
The purpose of this study is to evaluate the impact of auricular vagus nerve stimulation, applied in conjunction with an exercise treatment program, on pain and life quality in patients with Fibromyalgia Syndrome (FMS). To achieve the study objectives, 60 female patients between the ages 18 - 50, with diagnosed FMS according to American College of Rheumatology (ACR) 2010 diagnostic criteria, were randomly divided into 2 groups of 30. The first group was assigned 20 sessions of a home-based exercise program, while the second group was assigned 20 sessions of auricular vagus nerve stimulation and 20 sessions of a home-based exercise program. Patients were assessed before and after the treatments using the Visual Analog Scale (VAS) for pain, Beck Depression Scale for depression, Beck Anxiety Scale for anxiety, Fibromyalgia Impact Questionnaire (FIQ) for functional evaluation and Short Form-36 (SF-36) for life quality.

In this randomized controlled trial, comparisons within the groups revealed that both groups had statistically significant improvements in pain, depression, anxiety, functionality and life quality scores (p<0.05), whilst comparisons across the groups revealed that the group experiencing the vagus nerve stimulation had no statistically significant differences between the baseline scores, except for those of SF-36's sub-parameters of physical function, social functionality and pain. In fact comparisons across the groups after the interventions revealed that the group experiencing the vagus nerve stimulation had better scores but not statistically significant. From analysis of this data, the investigators observed that vagus nerve stimulation in FMS treatment did not give additional benefit together with exercise, except for three sub-parameters of SF-36. It was identified that further studies which separately investigate the effects of vagus nerve stimulation and exercise on FMS with longer follow-up periods and an increased number of patients are needed.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a syndrome, characterized by chronic widespread pain that continues for a minimum of 3 months and pain felt upon 11 out of 9 pairs of identified sore points. It is often accompanied by systemic symptoms such as fatigue, sleep disorders, cognitive dysfunction and depression . Moreover, headache, dysmenorrhea, irritable bowel syndrome, restless leg syndrome, chest pain, jaw pain, stomach ache, sensitive skin, mitral valve prolapses, Sicca symptoms, Raynaud phenomenon and female urethral syndrome accompany the clinical picture in many patients with FMS . This syndrome, the etiology of which is unknown, is commonly seen in women and the age of onset is usually 30 - 50 . Its prevalence among the general population is reported to be between 2.9 - 4.7 percent . While it is often seen in the adult population, it can also be observed in childhood or later age . Recent research studies show that various anomalies in genetic structure, autonomic nervous system (ANS), neurotransmitters, hypothalamic-hypophyseal-adrenal axe hormones, oxidative stress, pain modulation centers, central sensitization and muscular structure occur in FMS . The etiology of FMS is still not fully understood; nonetheless, the data reveals that this syndrome may stem from dysfunctionality in ANS . Sympathetic nervous system (SNS) dominance is widespread in FMS, chronic fatigue, irritable bowel syndrome and interstitial cystitis . A highly peripheral sympathetic tone causes regional ischemia, which in turn causes widespread pain. Therapeutic interventions that result in vasodilatation (e.g. exercise) and appropriate autonomic changes are proven to be effective for reducing pain levels .

The "great and perfect protector" of the body, the vagus nerve includes a neuro-endocrine-immune network that ensures homeostasis. The vagus nerve, which has reciprocal neural connections with more than one region of the brain, serves a control center that combines sensitive information and provides appropriate feedback responses. Recent studies show that the vagus nerve also encompasses inflammation, mood and pain regulation. All of these can be modulated with vagus nerve stimulation. Vagus nerve stimulation can generate a neuromodulating effect to activate other natural protective paths to improve health . The development of vagus nerve stimulation began in the 19th century. A number of new electrical stimulation devices have now been developed. Non-invasive transcutaneal devices stimulate the vagus nerve through the auricular branch or from the carotid. Moreover, they are used in the treatment of various disorders, such as epilepsy, pain and headache . Recent pre-clinical studies have shown that vagus nerve stimulation heavily modulates pain in humans and is quite effective. The use of a medical device allows the auricular branch of the vagus nerve to be stimulated without surgical intervention. Consequently, it has been found that the threshold of pain is elevated and mechanical pain sensitivity is reduced .

As a result of these completed studies, there is a possibility that FMS is a disease, which occurs through ANS impairment. Vagus nerve stimulation could be used as an additional treatment method to improve the ANS impairment. However, as there are no studies that investigate vagus nerve stimulation in FMS, this study is designed and executed.

MATERIAL AND METHOD

Our study, in which the researchers investigated the impact of auricular vagus nerve stimulation on pain and life quality in patients with FMS, was conducted in Beykoz Public Hospital's Department of Physiotherapy and Rehabilitation. A total of 60 female patients within the age range 18 - 50, with diagnosed FMS by a physiatrist according to 2010 ACR criteria, were included in this study. Only females were included to make groups homogenous and ended the age range at 50 to avoid comorbid illnesses seen in elderly people and also menopause. Pregnants, perimenopausal and postmenaopausal women are not included, also those experiencing any comorbid illnesses like neurological deficits, diabetes, neuropathic disorders, chronic inflammation, immune deficiency, cardiac disorders and current vitamin D intake were excluded from the study. In addition those who started using new drugs in the last month and during the study were not included. Patients who experienced vasovagal syncope in their past could not participate in the study.

Ethics committee approval was awarded by the Ethics Committee of Beykoz State Hospital Clinical Research prior to the commencement of the study. Written consent forms were obtained from all patients to demonstrate their consent to being included in the study. Patients were assessed twice during the study, firstly before treatment and then after treatment. Before the assessment, data was obtained from patients relating to age, height, weight, occupation, level of education, marital status, regular medication, general health complaints and the duration of these complaints. All responses were recorded. Patients were also asked to not participate in any other treatments during the study, in order to prevent any external influences on the data and study parameters.

Patients are diagnosed with FSM, in accordance with the ACR 2010 Diagnostic Criteria. A total of 60 patients are included in the study. Patients were randomly divided into two groups: an exercise (control) group and an exercise and vagus stimulation (treatment) group. Randomization was carried out by random number assignment. The exercise group began with 30 patients and the exercise and vagus stimulation group began with 30 patients. By the end of the study, there were 25 patients in the exercise group and 27 patients in the exercise and vagus stimulation group. Five patients in the exercise group were excluded as they had not completed the exercise program. 3 patients in the exercise and vagus stimulation group failed to complete the study and they missed treatment sessions. There was no blinding in the study.

The exercise group was assigned a program, which consisted of strengthening, stretching, isometric and posture exercises, targeting the body and upper and lower extremities. That program was home-based and the program was requested to be completed. Patients were asked to attend weekly face to face sessions with a total of 4 of these sessions in the study duration.

Patients in the exercise and vagus stimulation group received auricular vagus nerve stimulation at Beykoz Public Hospital's Department of Physical Therapy and Rehabilitation on 5 week days for 4 weeks, making up a total of 20 sessions with each session taking 30 minutes. Patients were admitted to the treatment as day visitors. Vagus nerve stimulation is carried out with a TENS device, which has specially designed surface electrodes in the shape of earphones, the size of which can be selected according to ear size. Electrodes were placed to correspond with the inner and rear surfaces of the tragus and the concha for both ears . The application is carried out, for 30 minutes, using a biphasic, asymmetrical waveform with a pulse duration that is less than 500 microseconds and a frequency of 10 Hertz. Amplitude is adjusted according to the sensory threshold level. Patients in this group were also assigned the same home-based exercise program assigned to the patients in the exercise group with application of the program 5 days a week with 2 sets per day and each set involved 10 repetitions of every exercise. Patients were asked to attend weekly face to face sessions with a total of 4 of these sessions in the study duration.

Measurements were performed twice, before and after the treatments. Patients were asked to complete the Turkish version of the Fibromyalgia Impact Questionnaire (FIQ), consisting of 21 questions, displaying the extent to which pain impacts the daily activities, social lives, moods and professional lives of the patients during the previous week.

Pain intensity was evaluated within the context of this study using the Visual Analog Scale (VAS). Patients were asked to select the corresponding interval for their own intensity of pain on a table of 0-100 mm with the explanation that 0 refers to no pain and 100 is excruciating pain .

Life quality of patients was evaluated using the SF-36 life quality scale. The Turkish validity and reliability of this scale was also carried out . Investigating life quality regarding overall health, this questionnaire contains 36 questions in 8 different categories .

The level of depression of patients was evaluated using the Beck Depression Scale. The Turkish validity and reliability of this scale was carried in 1988. It is a questionnaire that consists of 21 questions with 4 items and each item is awarded between 0-3 points (18).

The level of anxiety of patients was evaluated using the Beck Anxiety Scale.

Statistical Analysis

The presentation of variables acquired within the scope of the study such as sex, level of education and occupation includes numbers (n) and percentage values.

The Shapiro-Wilk test is used to determine whether the variables in the study are congruent with the normal distribution. Interquartile range (IQR) values for the variables without normal distribution and average±SD (Standard Deviation) values for the variables with normal distribution are provided in the descriptive statistics.

In the comparison of measurement values before and after the treatment, results of t-test for the variables with normal distribution and of Wilcoxon-Signed Rank test for the variables without normal distribution are provided.

In the comparison of treatment group and control group after the treatment, results of t-test for variables with normal distribution and of Mann Whitney-U test for variables without normal distribution are provided.

Chi-square and Likelihood Ratio Chi-Square tests were used to assess the relationship between patient and control group complaints, accompanying diseases, duration of pain and daily sports activities.

IBM SPSS Statistics 21.0 (IBM Corp. Released 2012. IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) and MS-Excel 2007 were used for statistical analyses and calculations. The level for statistical significance was accepted to be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Females 18- 50 of age

Exclusion Criteria:

* Pregnancy
* Menopause,
* Neurological deficits
* Diabetes
* Neuropathic disorders
* Chronic inflammation
* Immune deficiency
* Cardiac disorders
* Current drug usage
* Vasovagal syncope

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Short Form-36 Score | 4 weeks
  Life quality of patients was evaluated using the SF-36 life quality scale. The Turkish validity and reliability of this scale was carried out by Koçyiğit et al. Investigating life quality regarding overall health, this questionnaire contains 36 questions in 8 different categories.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.

CONTACTS AND LOCATIONS:
Overall Officials: kerem alptekin, Study Director — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wennemer HK, Borg-Stein J, Gomba L, Delaney B, Rothmund A, Barlow D, Breeze G, Thompson A. Functionally oriented rehabilitation program for patients with fibromyalgia: preliminary results. Am J Phys Med Rehabil. 2006 Aug;85(8):659-66. doi: 10.1097/01.phm.0000228677.46845.b2. PMID 16865020
- [Result] Gebre M, Woodbury A, Napadow V, Krishnamurthy V, Krishnamurthy LC, Sniecinski R, Crosson B. Functional Magnetic Resonance Imaging Evaluation of Auricular Percutaneous Electrical Neural Field Stimulation for Fibromyalgia: Protocol for a Feasibility Study. JMIR Res Protoc. 2018 Feb 6;7(2):e39. doi: 10.2196/resprot.8692. PMID 29410385
- [Result] Hamer HM, Bauer S. Lessons learned from transcutaneous vagus nerve stimulation (tVNS). Epilepsy Res. 2019 Jul;153:83-84. doi: 10.1016/j.eplepsyres.2019.02.015. Epub 2019 Feb 26. PMID 30952581
- [Result] Straube A, Ellrich J, Eren O, Blum B, Ruscheweyh R. Treatment of chronic migraine with transcutaneous stimulation of the auricular branch of the vagal nerve (auricular t-VNS): a randomized, monocentric clinical trial. J Headache Pain. 2015;16:543. doi: 10.1186/s10194-015-0543-3. Epub 2015 Jul 9. PMID 26156114

DOCUMENTS (1):
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT04260906/ICF_000.pdf